CLINICAL TRIAL: NCT02873481
Title: Centering Pregnancy Care + Yoga for Diverse Pregnant Women
Acronym: CPC+Y
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other); Southern Nursing Research Society (Unknown)
Responsible Party: Principal Investigator, Patricia Anne Kinser, Assistant Professor, Virginia Commonwealth University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20005136
Record Dates: First submitted 2016-04-05; First posted 2016-08-19 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Pregnancy
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (CPC+Y) (Experimental): Women in Centering Pregnancy Care (CPC) will receive the intervention which is a 30 minute yoga sessions during each of the 2-hour CPC meetings (CPC+Y)
  Interventions: Behavioral: Centering Pregnancy Care plus Yoga (CPC+Y)
- Comparison (CPC alone) (No Intervention): To strengthen our ability to examine causal relationships between the intervention and outcomes, we will use longitudinal comparison group data contributed from deidentified archival data from an existing IRB-approved study (PI: Masho) which includes pregnant women who participated in the CPC model of care alone (without the yoga component) and were followed throughout their pregnancies using numerous measures identical to those in the proposed study, including weight/BMI, depressive symptoms, anxiety, and stress.

INTERVENTIONS:
Behavioral: Centering Pregnancy Care plus Yoga (CPC+Y) — Gentle prenatal yoga for 30 minutes at the end of the Centering Pregnancy Care session
  Arms: Yoga (CPC+Y)

SUMMARY:
This is a pilot longitudinal mixed-methods study of pregnant women (n=20) who participate in CPC+Y at the VCU Health System Nelson Clinic or the Virginia Department of Health Richmond Health District's prenatal clinic (RHD) during their pregnancies. This pilot project will provide the necessary preliminary data to fuel an appropriately powered randomized controlled trial to evaluate the effects of CPC+Y in controlling weight gain, enhancing stress resilience, and improving maternal-child outcomes among overweight/obese diverse women. Because increasing physical activity has been found to have important mental health effects and maternal-child outcomes, it stands to reason that this innovative intervention has the potential to impact the way prenatal care is delivered in high risk populations.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women age 18 years or older
* currently participating in CPC at the VCU Health System Nelson Clinic or Richmond Health District

Exclusion Criteria:

* current physical conditions preventing participation in physical activity (ACOG guidelines: restrictive lung disease, hemodynamically significant heart disease, incompetent cervix, multiple gestation at risk of premature labor, persistent 2nd or 3rd trimester bleeding, placenta previa after 26 weeks gestation, premature labor, ruptured membranes, preeclampsia, severe anemia)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kinser, PhD, Principal Investigator — VCU
Locations (1):
- Virginia Commonwealth University School of Nursing, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yoga (CPC+Y) | Comparison (CPC Alone)
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga (CPC+Y) | Comparison (CPC Alone) | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (6.5) | 24.4 (5.6) | 26.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Retention/ Adherence
Description: Numbers of women who stayed in the study through their pregnancy and attended all intervention sessions
Time Frame: through study completion, an average of 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga (CPC+Y) | Comparison (CPC Alone)
Number analyzed (Participants) | 15 | 17
Participants | 15 | 17

2. Secondary Outcome: Self-efficacy for Physical Activity
Description: Physical Activity Self-Efficacy Scale (PASES): The Physical Activity Self-Efficacy Scale (PASES) is an 8 question scale which contains items about SM of physical activities and social support regarding PA. This psychometrically sound scale was selected because of its specific focus on SM of PA. Originally designed for adolescents, the wording has been slightly adapted for an adult sample. A higher score indicates higher levels of self-efficacy. Lowest possible score is 8; highest possible score is 40. Only participants in the intervention arm receive this particular instrument.
Time Frame: baseline (early pregnancy), end of pregnancy (approx 10 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga (CPC+Y)
Number analyzed (Participants) | 15
units on a scale
  Baseline | 25.8 (4.8)
  End of pregnancy | 25 (3.4)

3. Secondary Outcome: Salivary Biomarkers (α-amylase)
Description: salivary biomaker measure. This is an exploratory measure related to acute stress, yet it does not currently have known clinical associations with certain numeric levels of this measure (i.e., there is no identified "high" or "low" level of alpha-amylase). Only collected in the intervention group.
Time Frame: baseline (early pregnancy), mid-pregnancy (approx 4-5 months), end of pregnancy (approx 10 months)
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Yoga (CPC+Y)
Number analyzed (Participants) | 11
U/mL
  Baseline | 112.4145 (95.886)
  Mid-pregnancy | 99.59 (84.888)
  End of pregnancy | 127.045 (54.539)

4. Secondary Outcome: Depressive Symptoms
Description: Patient Health Questionnaire-9 (PHQ9): The PHQ-9 includes self-report items regarding depressive symptoms over the past two weeks. Total scores range from 0-27, where 0-4 indicates minimal depression, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately severe depressive symptoms, and ≥20 severe depressive symptoms.
Time Frame: baseline (early pregnancy), end of pregnancy (approx 10 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga (CPC+Y) | Comparison (CPC Alone)
Number analyzed (Participants) | 15 | 17
units on a scale
  Baseline | 5.2 (4.8) | 6.9 (5.3)
  End of pregnancy | 6.3 (5.9) | 12 (4.1)

5. Secondary Outcome: Stress
Description: Perceived Stress Scale (PSS): The Perceived Stress Scale-10 (PSS-10), a widely used, psychometrically sound instrument, will assess the degree to which a participant perceives stress in her life during the past month. The PSS-10 asks respondents to report about feelings such as unpredictability, uncontrollability, and overloading of stress in their lives; scores range from 0-40; higher scores correspond to a higher perceived stress level.
Time Frame: baseline (early pregnancy), end of pregnancy (approx 10 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga (CPC+Y) | Comparison (CPC Alone)
Number analyzed (Participants) | 15 | 17
units on a scale
  Baseline | 1.8 (2.2) | 1.3 (1.4)
  End of pregnancy | 0.33 (0.8) | 1.3 (1.4)

6. Secondary Outcome: Number of Subjects Participating in Focus Group
Description: Women will volunteer to discuss their experiences (acceptability) with the intervention through focus groups conducted following the intervention period
Time Frame: at intervention completion, an average of 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga (CPC+Y)
Number analyzed (Participants) | 8
Participants | 8

7. Secondary Outcome: Recruitment Feasibility
Description: Numbers of women who agreed to participate in the study;
Time Frame: at intervention completion, an average of 20 weeks
Measure: Number; unit: participants
Arm/Group | Yoga (CPC+Y) | Comparison (CPC Alone)
Number analyzed (Participants) | 15 | 17
participants | 15 | 17

ADVERSE EVENTS:
Time Frame: intervention period (9 months)
Arm/Group | Yoga (CPC+Y) | Comparison (CPC Alone)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No